CLINICAL TRIAL: NCT01214993
Title: A Phase 1, Open Label, Placebo-Controlled Study to Evaluate the Effect of GSK1349572 on Iohexol and Para-Aminohippurate Clearance in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Shionogi (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 114819
Record Dates: First submitted 2010-10-01; First posted 2010-10-05 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Infections, Human Immunodeficiency Virus and Tuberculosis
Keywords: GSK1349572; para-aminohippurate; iohexol
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; Tuberculosis | interventions — dolutegravir; Iohexol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): There will be a screening visit within 30 days prior to the first dose of study drug. In this treatment arm, all subjects will receive GSK1349572 50mg (two 25mg tablets) q24h for 14 days. Subjects will also receive iohexol and PAH infusions on Days -1, 7 and 14. There will be a follow-up visit 7-10 days after the last dose of study medication.
  Interventions: Drug: GSK1349572; Drug: Iohexol Injection; Drug: Para-aminohippurate infusion
- Treatment B (Experimental): There will be a screening visit within 30 days prior to the first dose of study drug. In this treatment arm, all subjects will receive GSK1349572 50mg (two 25mg tablets) q12h for 14 days. Subjects will also receive iohexol and PAH infusions on Days -1, 7 and 14. There will be a follow-up visit 7-10 days after the last dose of study medication.
  Interventions: Drug: GSK1349572; Drug: Iohexol Injection; Drug: Para-aminohippurate infusion
- Treatment C (Placebo Comparator): There will be a screening visit within 30 days prior to the first dose of study drug. In this treatment arm, all subjects will receive placebo q24h for 14 days. Subjects will also receive iohexol and PAH infusions on Days -1, 7 and 14. There will be a follow-up visit 7-10 days after the last dose of study medication.
  Interventions: Drug: Placebo; Drug: Iohexol Injection; Drug: Para-aminohippurate infusion

INTERVENTIONS:
Drug: GSK1349572 — GSK1349572 is an experimental drug in the integrase inhibitor class of drugs to treat human immunodeficiency virus (HIV)
  Arms: Treatment A; Treatment B
Drug: Placebo — Placebo is a tablet with no drug in it.
  Arms: Treatment C
Drug: Iohexol Injection — Iohexol is an FDA approved radiologic contrast medium
  Other Names: OMNIPAQUE
Drug: Para-aminohippurate infusion — Para-aminohippurate is an agent to measure effective renal plasma flow.

SUMMARY:
The current study is designed to confirm the mechanism behind the increase in serum creatinine observed during GSK1349572 therapy; specifically, the study will determine whether GSK1349572 has any effect on glomerular filtration rate (GFR) or effective renal plasma flow. Absent such effects, one may conclude that the small increases in serum creatinine observed are due to the inhibition of the tubular secretion of creatinine via organic cation transporter 2 (OCT2) consistent with in vitro data. .

DETAILED DESCRIPTION:
GSK1349572 is an integrase inhibitor being developed for the treatment of human immunodeficiency virus (HIV)-1 infection by GlaxoSmithKline (GSK) on behalf of Shionogi-ViiV Healthcare LLC. In healthy subjects and in dose-ranging clinical trials of GSK1349572, subjects showed a small, reversible increase in serum creatinine concentrations as compared to the control groups; this occurred early during study drug administration and did not progress over time. In vitro data demonstrate that GSK1349572 inhibits the organic cation transporter (OCT2), which mediates the tubular secretion of creatinine; drugs such as cimetidine with similar effects on OCT2 lead to a nonpathological increase in creatinine with no effect on glomerular filtration rate (GFR). The current study is designed to confirm the mechanism behind the increase in serum creatinine observed during GSK1349572 therapy; specifically, the study will determine whether GSK1349572 has any effect on GFR or effective renal plasma flow. Absent such effects, one may conclude that the small increases in serum creatinine observed are due to the inhibition of the tubular secretion of creatinine via OCT2.

Subjects will be given GSK1349572 50mg once daily, 50mg twice daily or placebo once daily for 14 days. Changes in the subject's GFR will be measured through administration of iohexol and effective renal plasma flow will be measured using Para-Aminohippurate (PAH) on days -1, 7 and 14. Changes in serum creatinine and other renal biomarkers will be evaluated at baseline and at various time points throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with normal renal function defined as creatinine clearance greater than or equal to 80 mL/min/1.73m2 measured by 24 urine collection
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase and bilirubin less than or equal to 1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<147 pmol/L) is confirmatory]. OR Child-bearing potential and agrees to use one of the contraception methods listed in the protocol for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the follow-up visit.
* Body weight greater than or equal to 50 kg for males and 45 kg for females and body mass index (BMI) within the range 18.5- 31.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* History of sensitivity to any of the study medications, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation. A subject with any history of allergic reaction to contrast media should not be enrolled.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* If heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 drinks/week for men or >7 drinks/week for women. One drink is equivalent to (12 g alcohol) = 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* Has a history or regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
* Pregnant females as determined by positive serum or urine human chorionic gonadotrophin (hCG) test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy, peptic ulceration, inflammatory bowel disease or pancreatitis should be excluded.
* History/evidence of clinically significant pulmonary disease.
* History of significant renal or hepatobiliary diseases. Subjects with a history of nephrolithiasis will be excluded.
* Any subject with evidence of microalbuminuria at screening defined as albumin-to-creatinine ratio in a random spot urine ≥ 0.03 mg/mg OR 30 mg/g.
* History of severe or serious psychiatric disease ever requiring hospitalization, history of suicidal ideation or suicidal attempt, or undergoing psychiatric treatment will be excluded from study participation.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* History of Gilbert's disease.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects.
* Exclusion criteria for screening ECG per protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Glomerular Filtration Rate (GFR) as measured by iohexol plasma clearance at days -1, 7 and 14 | 14 days

SECONDARY OUTCOMES:
Serum creatinine, creatinine clearance (CrCL) as measured by 24-hour urine collection, and extra-glomerular creatinine excretion (EGCE) at days -1, 7, 14 and follow-up | 24 days
Serum concentrations of Cystatin-C, 24-hour urinary excretions of albumin, total protein, beta2-microblobulin, N-acetyl-beta-d-glucosaminidase (NAG) and retinol binding protein at days -1, 7, 14 and at follow-up | 24 days
Effective renal plasma flow (ERPF) as measured by plasma clearance of Para Aminohippurate (PAH) at days -1, 7 and 14 | 14 days
Safety and tolerability parameters, including adverse event, concurrent medication, clinical laboratory and vital signs assessments. | 24 days
Day 14 GSK1349572 PK parameters including area under the concentration curve (AUC)(0-tau), AUC(0-24), concentration (C)max, C0, and Ctau. | day 14

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Minneapolis, Minnesota, United States